CLINICAL TRIAL: NCT05586386
Title: Effect of Dark Sweet Cherry (DSC) Supplementation on the Gut Microbiota-liver-brain Axis in Obese Adults
Brief Title: Cherries Role in Gut Microbiota-liver-brain Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Texas A&M University (Other)
Responsible Party: Principal Investigator, Giuliana Noratto, Research Associate Scientist, Texas A&M University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB2019-0597F
Record Dates: First submitted 2022-10-04; First posted 2022-10-19 (Actual); Last update posted 2022-10-19 (Actual); Status verified 2022-10

CONDITIONS: Obesity
Keywords: dark sweet cherry; anthocyanins; obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Intervention Model Description: Group 1: Obese adults (BMI: 30-40): 200 mL (~6.7 oz.) of dark sweet cherry (DSC) juice supplemented with 3g of DSC powder twice per day for 30 days.
  Group 2: Obese adults (BMI: 30-40): 200 mL (~6.7 oz.) of placebo juice twice per day for 30 days.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cherry group (Experimental): Obese adults were asked to consume 200 mL of DSC juice supplemented with 3g of DSC powder twice / day for 30 days.
  Interventions: Other: Cherry group
- Placebo group (Experimental): Obese adults were asked to consume 200 mL of placebo juice supplemented twice / day for 30 days.
  Interventions: Other: Placebo group

INTERVENTIONS:
Other: Cherry group — 200 mL of DSC juice twice/day supplemented with 3g of DSC powder twice/day for 30 days
  Arms: Cherry group
Other: Placebo group — 200 mL of placebo juice twice/day
  Arms: Placebo group

SUMMARY:
Sweet cherries (Prunus avium) are a good source of bioactive compounds including dietary fiber and phytochemicals which have been credited with multiple health benefits, including anti-inflammatory and antioxidant properties as well as preventing obesity-related metabolic disorders. However, most studies have shown such benefits using in vitro or animal models. The aim of this study was to examine the influence of DSC consumption on obesity-associated inflammation, metabolic disorders, cognitive impairment, and gut dysbiosis in obese individuals.

DETAILED DESCRIPTION:
The duration of an individual's participation in the study was 45 days (15 days for the run-in period plus 30 days of intervention):

* Screening: Eligible participants were contacted through e-mail and invited to participate in a familiarization session in which detailed information about the study along with the consent statement form was presented. Participants who met the eligibility criteria and signed the consent were scheduled for screening visits. During the screening visits, the anthropometric (waist circumference, height, weight, and BMI) and wellness measurements (blood pressure, heart rate, and oxygen saturation) were measured.
* Run-in period: Participants were asked to complete a 2-week run-in period in which dietary supplements were removed from the diet while maintaining usual dietary patterns. During the run-in period, participants were asked to complete 24-hour dietary records for 5 days to have the baseline information related to their dietary patterns. In addition, participants were asked to reduce their intake of polyphenol and fiber-rich foods. After the completion of the 2-week run-in period, participants were allocated into cherry or placebo groups according to BMI, age, and gender and scheduled for study visits 1, 15, and 30.
* Intervention: During the 30-day cherry or placebo supplementation, participants were asked to maintain usual physical activity and diet, and to minimize the intake of foods high in polyphenol content. Nutritional habits were evaluated using 15-day dietary records collected on Myfitnesspal. Participants were instructed to drink a cherry juice or corresponding placebo twice a day for 30 days. At each study visit (study days 1, 15, and 30), wellness checks (blood pressure, heart rate, and oxygen saturation) and anthropometric measurements (body weight, height, % of body fat, body mass index (BMI), waist and hip circumference) were recorded. Biomarkers of inflammation, metabolic disorders, and liver health were assessed on blood samples collected on study days 1 and 30. Participants were instructed to fast for 12 h. before each study appointment and to drink plenty of water to facilitate blood draws. Blood fractions were aliquoted and stored at -80 C until analyses. The gut microbiota composition was assessed on stool samples collected on study days 1 and 30. Participants were given stool collection kits and instructed to avoid the use of laxatives, stool softeners, and antiacids within 48 hr. before stool collection. Participants were asked to bring their samples on study days 1 and 30 within 2 h. of collection or to freeze them if collected a day prior until transport to our facility. Stool samples received by the research personnel were immediately stored at -80 ⁰C until analysis. Intestinal permeability, which is a feature of intestinal barrier function, was evaluated through the lactulose/mannitol/sucralose test in urine samples collected on study days 1 and 30. This test was optional for participants. On study days 1 and 30, participants were given urine collection kits and instructed to collect their samples within 5 h of drinking a sugary solution containing lactulose, mannitol, and sucralose. Samples were stored at -20°C until analysis. Cognitive function was monitored on study days 1 and 30 through interviewer-administered tests that provided information on executive function skills (visual search, scanning, working memory, processing speed, and attention). In addition, visual cognitive performance was monitored during the last 15 days of the intervention using the Visual Cognitive Testing and Training: NeuroTracker™ CORE program (NT) from CogniSens Inc, which is a single-task integrative perceptual-cognitive training system.

ELIGIBILITY:
Inclusion Criteria:

* Male or female at least 18 years old;
* No history of chronic diseases or intestinal disorders.
* BMI: ≥ 30 and ≤ 40.

Exclusion Criteria:

* History of acute cardiac event, stroke, or cancer
* Alcohol or substance abuse within the last 6 months
* Recurrent admittance to the hospital (twice or more)
* Allergy, intolerance, or sensitivity to berries
* Hepatitis (B or C) or HIV
* Smoking more than 1 pack/week
* Liver or renal dysfunction
* Diabetic retinopathy
* History of glaucoma, retinitis pigmentosa, optic neuropathy, retinal vascular occlusions, strabismus, macular degeneration or autoimmune disorders related to visual health
* History of dizziness/fainting during and after blood draws
* Known lactose intolerance, gluten sensitivity, or celiac disease
* Currently on medications/antibiotics
* Pregnancy or lactation (or planned pregnancy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-02-06 (Actual); Primary Completion 2021-09-20 (Actual); Study Completion 2021-09-20 (Actual)

PRIMARY OUTCOMES:
Change from baseline intestinal microbiota composition at 30 days | At day 1 (baseline) and day 30
  16S rRNA sequencing was used to evaluate the intestinal microbiota composition in stool samples collected on day 1 (baseline) and 30.
Change from baseline liver health biomarkers at 30 days | At day 1 (baseline) and day 30
  Liver enzymes (alanine aminotransferase (ALT), aspartate aminotransferase (AST), and alkaline phosphatase) levels were measured on fasting blood samples collected on day 1 and 30.
Change from cognitive function at 30 days | At day 1 (baseline) and day 30
  The trail making tests (A and B) were administered on day 1 and 30 to evaluate executive attention, and visual-spatial functions (visual search and scanning, sequencing).
Change from cognitive function at 30 days | At day 1 (baseline) and day 30
  The Digit Span tests (Forward and Backward) were administered on day 1 and 30 to evaluate working memory and concentration skills.
Change from cognitive function at 30 days | At day 1 (baseline) and day 30
  The Digit Span Substitution test was administered on days 1 and 30 to evaluate processing speed, sustained attention, and visual perception.

SECONDARY OUTCOMES:
Change from baseline inflammatory biomarkers at 30 days | At day 1 (baseline) and day 30.
  Biomarkers of inflammation such as pro-inflammatory cytokines (interleukins IL-6, -1β, -8, interferon gamma (INFγ), and monocyte chemoattractant (MCP-1)), and C-reactive protein (CRP) were assessed on fasting blood samples collected on day 1 (baseline) and day 30.
Visual cognitive performance | From day 15 to day 30.
  The visual cognitive testing and training: NeuroTracker (NT)™ CORE program was used to evaluate attention (sustained, selective, divided, inhibition), memory (short-term and working) and information processing speed. Participants completed ten sessions between days 15 and 30.
Change from baseline lipid profile biomarkers at 30 days | At day 1 (baseline) and day 30
  Cholesterol (HDL, LDL, non-HDL) and triglyceride levels were measured on fasting blood samples collected on day 1 (baseline) and day 30.

CONTACTS AND LOCATIONS:
Locations (1):
- Texas A&M University, College Station, Texas, United States